CLINICAL TRIAL: NCT04092660
Title: Intervention to Enhance Adherence to Mandibular Advancement Appliance in Patients With Obstructive Sleep Apnoea: A Randomized Control Trial
Brief Title: Increasing the Use of an Anti-snoring Mouth Guard (Mandibular Advancement Appliance) to Prevent Upper Airway Collapse During Sleep in Patients With Obstructive Sleep Apnoea.
Acronym: IPOSAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 262092
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Multicentre Randomized Control Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Care Group (Experimental): The Intervention care group will receive the Mandibular Advancement Appliance (MAA) or the anti-snoring mouthguard. Additionally, they will also receive special support in the form of behaviour change interventions. The behavior change interventions consist of motivational interviewing, will be shown a video highlighting the negative consequences of sleep apnoea.
  Booster calls at week 3,6, 18 and 12 for verbal encouragement and to resolve any technical problems with the device.
  Participants will be asked to complete questionnaires regarding their personality, socio-economic status, social support and quality of sleep and life.
  Interventions: Behavioral: Behaviour change Intervention Based on Health Action Process Approach Model; Device: Mandibular Advancement Appliance (MAA) or Anti-snoring mouth guard
- Standardized Care Group (Active Comparator): The standardized care group will only receive the Mandibular Advancement Appliance (MAA) or the anti-snoring mouthguard along with routine care and will be called for follow up at 3rd and 6th month of treatment to assess their use and to resolve any technical problems with the device.
  Participants will be asked to complete questionnaires regarding their personality, socio-economic status, social support and quality of sleep and life at the initial visit and subsequent follow-up.
  Interventions: Device: Mandibular Advancement Appliance (MAA) or Anti-snoring mouth guard

INTERVENTIONS:
Behavioral: Behaviour change Intervention Based on Health Action Process Approach Model — The Behaviour change intervention based on the Health Action Process Approach model entails delivering interventions in a staged manner. Following are the intervention that will be delivered along with the time point of the delivery.
  1. Health Pamphlet at the initial screening
  2. Sleep Apnoea video highlighting the negative consequences at the day of the fitting of the appliance
  3. Counseling involving motivational interviewing for both the participant and the participant's partner at the day of fitting of the appliance and follow up visits.
  4. Booster phone calls in between the follow-up visits
  Arms: Intervention Care Group
Device: Mandibular Advancement Appliance (MAA) or Anti-snoring mouth guard — Patients with mild-to-moderate sleep apnoea are treated with Mandibular Advancement Appliances [MAA] also known as Anti-snoring mouth guards or Oral appliances. These are best made to fit and use the teeth to hold them in place during sleep. They work by moving (in a gradual fashion) the bottom jaw forward, opening the airway at the back of the throat.
  Both the arms- Intervention arm and Standardized arm will be given the anti-snoring mouth guard. The usage of the device will be measured subjectively by providing a sleep diary to the participants to record the hour of the usage and objectively by downloading the data from a micro sensor chip embedded in the device.

SUMMARY:
Obstructive Sleep Apnoea (OSA) is a sleep-related breathing disorder that is characterized by the repeated collapse of the upper airway during sleep, resulting in sleep deprivation. Mandibular Advancement Appliances (MAA) or Oral Appliances (OA) is prescribed for the patients with OSA and they have been shown to be effective. However, they rely entirely on the patient's acceptance and use. The aim of this study is to assess whether interventions- additional support approaches, will help patients use their MAA more as compared to those who receive routine care.

The investigators also will try and identify factors that help us to understand why some patients choose to wear the MAA more than others. Adults (≥40 years) with a confirmed diagnosis of OSA (apnoea-hypopnoea index >5) and referred for MAA therapy will be included in this study. It is a multicentre study comprised of recruiting patients from secondary care. Patients will be provided with information in relation to the study and written informed consent obtained at their subsequent appointment for placement of MAA.

Patients will be randomly assigned to Intervention Care (IC) and Standardised care (SC). Patients will also be provided with a sleep diary to subjectively record their hours of sleep and usage of MAA and an objective adherence record from the micro-sensor included in their MAA design. Data indicating adherence will be collected and evaluated, both subjectively at 3- (T2) and 6-months (T3) and objectively by downloading the data stored within a micro-sensor placed in the MAA device. At the end of the follow-up, the investigators also plan to undertake a qualitative one-to-one interview with patients compliant (users) and non-compliant (non-users) to identify their views of what helps and/or prevents their adherence.

DETAILED DESCRIPTION:
The present study aims to assess whether special support approaches i.e. Interventions influence patients with Obstructive sleep apnoea (OSA), to use the Mandibular Advancement Appliance (MAA) or the anti-snoring mouth guard, more as compared to those who receive standard care.

Factors such as mood, anxiety, stress, depression, socioeconomic status, and social support play an important role in the ability of the patients to make decisions about using the appliance. Thus, the investigators also aim to explore the potential role these factors play in the decision-making process to help future patients make most of their treatments.

Patients meeting the selection criteria will be provided with a patient information leaflet, explaining the whole study. Interested patients will be asked to sign the Informed Consent, after which they will be randomly assigned into two groups- Intervention Care group (IC) and Standardized Care group (SCG).

Patients will be provided with a sleep diary to record their hours of sleep and usage of MAA, which will give a subjective record of the adherence (duration of usage of MAA) and an objective record of the adherence will be collected from a sensor present in the MAA.

At Initial Screening, the patient's age, gender, body mass index (BMI) and neck circumference will be recorded. Patients in the IC group will receive a Health Pamphlet about OSA, specially designed for this study. The IC group's knowledge of OSA will be assessed along with their partner's. Patients in the IC group will be shown a 10 min video highlighting the negative impact of OSA. While patients in the SC group will only be provided with a pamphlet about OSA and MAA as per standard routine care.

Patients of both the group will be asked to complete questionnaires regarding their personality, socioeconomic status, social support and quality of sleep and life.

Along the course of the treatment, patients in the IC group will be contacted by telephone at 3, 6, 18, and 21 weeks into the treatment to solve any technical problems with the appliance and for verbal encouragement.

Both IC and SC groups will be called for follow-up at 3 and 6 months into the treatment. Data indicating the hours of usage of the MAA will be collected at 3 and 6 months to assess whether patients in the IC group wore the appliance for more hours as compared to those who are in the SC group. Patients will also be required to complete questionnaires at follow-up appointments. Data from the questionnaires will be analyzed to identify the factors influencing patients adherence to MAA.

At the end of follow-up, one-to-one interviews will be conducted with both (n=5-10) compliant (users) and non-compliant (non-users) patients. It will comprise of questions, which will address the following topics:

* Patient's awareness of risks and benefits of OSA
* Barriers and Facilitators of MAA therapy The interviews will be conducted face-to-face and will be recorded using an audio recorder device and transcribed by a third party, Essential Secretary LTD.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 40 years old)
* Confirmed diagnosis of OSA (AHI ≥ 5)
* Referred for MAA therapy
* Must be able to understand, read and write English; with the assistance of a translator

Exclusion Criteria:

* Insufficient teeth for MAA fabrication
* Poor dental and/or periodontal health
* Symptomatic Temporomandibular Disorder (TMD)
* Previously used an MAA
* Patients with Epilepsy

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2019-12-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Adherence- the number of hours the patient uses the MAA or anti-snoring mouth guard every night | 3 months
  the number of the hours the patient uses the appliance every night will be measured both objectively and subjectively at 3 and 6 months to assess the effectiveness of the interventions in enhancing adherence to MAA.
Adherence-the number of hours the patient uses the MAA or anti-snoring mouth guard | 6 month
  the number of the hours the patient uses the appliance every night will be measured both objectively and subjectively at 3 and 6 months to assess the effectiveness of the interventions in enhancing adherence to MAA.

SECONDARY OUTCOMES:
Self-efficacy, risk perception, outcome expectancy | Initial screening, 3 and 6 month
  Self-efficacy, risk perception, outcome expectancy will be measured using the Self-efficacy Measure for Sleep Apnoea (SEMSA) questionnaire
Socio-economic status | Initial Screening
  Socio-economic Status questionnaire based on National Statistics Socio-Economic Classification.
Social support | Initial Screening
  Social Support Questionnaire
Sleep Quality | Initial Screening and 6 month
  Sleep Quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire
Sleepiness Score: How likely is the participant to fall asleep in certain situations? | Initial Screening and 6 month
  Epworth Sleepiness Scale Questionnaire will be used to assess the sleepiness score.
Health related Quality of Life | Initial Screening and 6 month
  EQ-5D questionnaire will be used to measure the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ama Johal, Study Chair — Queen Mary University of London
Locations (1):
- Royal London Dental Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tallamraju H, Newton JT, Fleming PS, Johal A. Intervention to enhance adherence to mandibular advancement appliance in patients with obstructive sleep apnoea: study protocol for a randomised clinical trial. Trials. 2021 Oct 13;22(1):699. doi: 10.1186/s13063-021-05582-1. PMID 34645490